CLINICAL TRIAL: NCT01836445
Title: Efficacy of Internet-based HIV Prevention
Brief Title: Keep It Up! 2.0: A Comparison of Two Online HIV Intervention Programs for Young Men Who Have Sex With Men
Acronym: KIU!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Emory University (Other); Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Brian Mustanski, Associate Professor, Department of Medical Social Sciences; Director, IMPACT Program, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01DA035145-01 (NIH); 1R01DA035145-01 (NIH)
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: HIV; Gonorrhea; Chlamydia
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Keep It Up! Intervention (Experimental): The KIU! intervention is a multi-media online HIV prevention program developed specifically for young (18-29 years old) men who have sex with men (MSM) who recently tested HIV negative. Intervention content includes discussions of community involvement, scenarios on hooking-up online, communication skills in relationships (including negotiating safer sex), condom use, HIV knowledge, and HIV/STI risks. Information is presented in various formats like games, animation, and videos to address gaps in HIV knowledge, motivate safer behaviors, teach behavioral skills, and instill self-efficacy for preventive behaviors. The intervention is completed across three sessions, done at least 24 hours apart (i.e. at least 3 days), and takes about 2 hours total to complete.
  Interventions: Behavioral: Keep It Up!
- HIV Knowledge Control (Active Comparator): The control condition reflects HIV information that is currently available on many websites so as to understand how the KIU! intervention improves upon what is currently available online. It is not tailored to YMSM, non-interactive, and focused on HIV/STI knowledge. The control is completed across three sessions done at least 24 hours apart (i.e. at least 3 days).
  Interventions: Behavioral: HIV Knowledge Control

INTERVENTIONS:
Behavioral: Keep It Up!
  Other Names: KIU!; KIU! 2.0; Keep It Up! 2.0
  Arms: Keep It Up! Intervention
Behavioral: HIV Knowledge Control
  Arms: HIV Knowledge Control

SUMMARY:
Young men who have sex with men (YMSM) account for almost 70% of HIV diagnoses among all young people in the U.S. and are alone in facing an increasing rate of infections. Because YMSM are less likely to receive relevant sexual health education in traditional settings (e.g. schools, community), the Internet is a unique route of reaching and helping YMSM.

The purpose of this study is to compare two different versions of an online HIV prevention program for YMSM. The study is being conducted by researchers at Northwestern University in Chicago, Hunter College in New York City, and Emory University in Atlanta. A total of 900 YMSM will be enrolled into this study from the clinics of community partners in Chicago, New York, and Atlanta.

Participants will be randomly assigned to one of two versions of the program. Some topics in the program include HIV facts and myths, sexually transmitted infections (STIs), and condom use. All participants, regardless of the program version they receive, will also take at-home urine and rectal tests for the STIs chlamydia and gonorrhea. After completing the program, participants will be contacted three more times over the course of a year for follow-up sessions and surveys.

The research team hypothesizes that the YMSM-specific prevention program will lead to a significant reduction in the frequency of unprotected anal sex acts and new STI infections compared to the HIV knowledge program that is for a general audience. The YMSM-specific program will also lead to improvements in secondary knowledge, motivation, and skills outcomes.

In order for the research team to measure the effectiveness of the YMSM-specific prevention program and determine if the study hypothesis is correct, participants will be asked questions about themselves, including questions about their sexual orientation, sexual experiences, health practices, including drug use, health knowledge, and questions about their feelings and emotions. Based on this information, the research team hopes to later change, improve, or expand the program to better address the needs of YMSM.

ELIGIBILITY:
Inclusion Criteria:

* Birth male who identifies as male and reports sexual contact with another male
* Received an HIV negative test result from a participating clinic/recruitment site
* Unprotected anal sex with another male in the last 6 months
* Ability to read English at 8th grade level

Exclusion Criteria:

* HIV positive
* Female or Transgender
* No email address for contact
* Currently in a monogamous relationship lasting longer than 6 months
* Participated in previous versions of KIU!

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 901 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mustanski, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Hunter College, New York, New York

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). HIV Surveillance in Adolescents and Young Adults. 2010.
- [Background] Centers for Disease Control and Prevention (CDC). Trends in HIV/AIDS diagnoses among men who have sex with men--33 states, 2001-2006. MMWR Morb Mortal Wkly Rep. 2008 Jun 27;57(25):681-6. PMID 18583954
- [Background] Prejean J, Song R, Hernandez A, Ziebell R, Green T, Walker F, Lin LS, An Q, Mermin J, Lansky A, Hall HI; HIV Incidence Surveillance Group. Estimated HIV incidence in the United States, 2006-2009. PLoS One. 2011;6(8):e17502. doi: 10.1371/journal.pone.0017502. Epub 2011 Aug 3. PMID 21826193
- [Background] Mustanski B, Lyons T, Garcia SC. Internet use and sexual health of young men who have sex with men: a mixed-methods study. Arch Sex Behav. 2011 Apr;40(2):289-300. doi: 10.1007/s10508-009-9596-1. Epub 2010 Feb 25. PMID 20182787
- [Derived] Mustanski B, Parsons JT, Sullivan PS, Madkins K, Rosenberg E, Swann G. Biomedical and Behavioral Outcomes of Keep It Up!: An eHealth HIV Prevention Program RCT. Am J Prev Med. 2018 Aug;55(2):151-158. doi: 10.1016/j.amepre.2018.04.026. Epub 2018 Jun 28. PMID 29937115
- [Derived] Mustanski B, Madkins K, Greene GJ, Parsons JT, Johnson BA, Sullivan P, Bass M, Abel R. Internet-Based HIV Prevention With At-Home Sexually Transmitted Infection Testing for Young Men Having Sex With Men: Study Protocol of a Randomized Controlled Trial of Keep It Up! 2.0. JMIR Res Protoc. 2017 Jan 7;6(1):e1. doi: 10.2196/resprot.5740. PMID 28062389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2013 to December 2015, 901 participants were recruited and enrolled from (1) community-based HIV testing organizations in Atlanta, Chicago, and New York; (2) local health department clinics in Chicago; (3) street outreach in Atlanta, Chicago, and New York; and (4) local and national advertising.
Pre-assignment Details: Participants were randomized after completing a baseline assessment and STI testing.
Groups:
- Keep It Up! Intervention: The KIU! intervention is a multi-media online HIV prevention program developed specifically for young (18-29 years old) men who have sex with men (MSM) who recently tested HIV negative. Intervention content includes discussions of community involvement, scenarios on hooking-up online, communication skills in relationships (including negotiating safer sex), condom use, HIV knowledge, and HIV/STI risks. Information is presented in various formats like games, animation, and videos to address gaps in HIV knowledge, motivate safer behaviors, teach behavioral skills, and instill self-efficacy for preventive behaviors. The intervention is completed across three sessions, done at least 24 hours apart (i.e. at least 3 days), and takes about 2 hours total to complete.
  Keep It Up!
- HIV Knowledge Control: The control condition reflects HIV information that is currently available on many websites so as to understand how the KIU! intervention improves upon what is currently available online. It is not tailored to YMSM, non-interactive, and focused on HIV/STI knowledge. The control is completed across three sessions done at least 24 hours apart (i.e. at least 3 days).
  HIV Knowledge Control
Period: Intervention Modules
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Started | 445 | 456
Completed | 375 | 434
Not Completed | 70 | 22
Period: 3 Month Follow-up Assessment
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Started | 445 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention) | 456 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention)
Completed | 348 | 409
Not Completed | 97 | 47
Period: 6 Month Follow-up Assessment
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Started | 445 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention) | 455 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention)
Completed | 342 | 380
Not Completed | 103 | 75
Period: 12 Month Follow-up Assessment
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Started | 445 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention) | 455 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention)
Completed | 370 | 391
Not Completed | 75 | 64
Period: 12 Month STI Testing
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Started | 445 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention) | 455 (All enrolled participants allowed to complete follow-up regardless of if they completed intervention)
Completed | 365 | 378
Not Completed | 80 | 77

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control | Total
Number analyzed (Participants) | 445 | 456 | 901
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.27 (3.02) | 24.15 (2.89) | 24.21 (2.95)
Age, Customized [Count of Participants; unit: Participants]
  18 - 24 | 233 | 244 | 477
  25 - 29 | 211 | 212 | 423
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 445 | 456 | 901
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American | 1 | 4 | 5
  Asian | 15 | 22 | 37
  Black or African American | 106 | 113 | 219
  Hispanic or Latino | 135 | 125 | 260
  White | 165 | 165 | 330
  More than one race | 15 | 17 | 32
  Unknown or Not Reported | 8 | 10 | 18
Condomless Anal Sex [Mean (Standard Deviation); unit: condomless anal sex acts] | 4.3 (13.1) | 3.4 (6.7) | 3.9 (9.9)
Sexually Transmitted Infections [Count of Participants; unit: Participants] — Enrolled participants who returned STI test kits for analysis at Baseline (n = 896) Population: Enrolled participants who returned STI test kits for analysis at baseline. Denominator varies by testing site and study arm: urethral (control - 452; intervention - 441) rectal (control - 449; intervention - 442)
  Participants
    Urethral Chlamydia: number analyzed (Participants) | 441 | 452 | 893
    Urethral Chlamydia | 15 | 7 | 22
    Urethral Gonorrhea: number analyzed (Participants) | 441 | 452 | 893
    Urethral Gonorrhea | 3 | 4 | 7
    Rectal Chlamydia: number analyzed (Participants) | 442 | 449 | 891
    Rectal Chlamydia | 47 | 30 | 77
    Rectal Gonorrhea: number analyzed (Participants) | 442 | 449 | 891
    Rectal Gonorrhea | 29 | 16 | 45
    Any STI: number analyzed (Participants) | 443 | 453 | 896
    Any STI | 82 | 50 | 132
Education [Count of Participants; unit: Participants] — Enrolled participants who completed questions on educational background at baseline
  Participants
    Junior High School | 0 | 1 | 1
    Partial High School | 10 | 7 | 17
    High School Graduate/GED | 60 | 35 | 95
    Partial College (at Least One Year) | 116 | 136 | 252
    College Education | 203 | 215 | 418
    Graduate Degree | 56 | 62 | 118
Employment [Count of Participants; unit: Participants] — Enrolled participants who were employed and answered follow-up questions on employment status at baseline Population: Only participants who were employed and answered the follow-up questions on employment are included in the analysis population.
  Participants
    number analyzed (Participants) | 338 | 363 | 701
    Full Time | 223 | 228 | 451
    Part Time | 115 | 135 | 250

OUTCOME MEASURES:

1. Primary Outcome: Participants Self-Reporting Condomless Anal Sex at Baseline and 3 Months
Description: Change in self-report of condomless anal sex acts at three months.
Time Frame: Baseline, 3 Months
Population: Enrolled participants who completed assessments on their sexual risk behaviors (e.g. condomless anal sex (CAS) acts) at baseline and 3 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 445 | 454
Participants
  Baseline | 304 | 312
  3 Month Follow-up: number analyzed (Participants) | 362 | 406
  3 Month Follow-up | 148 | 184
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Superiority; p = 0.20, Regression, Logistic; Prevalence Ratio = 0.90, 95% CI 2-sided [0.76 to 1.06]

2. Primary Outcome: Participants Self-Reporting Condomless Anal Sex at Baseline and 6 Months
Description: Change in self-report of condomless anal sex acts at six months.
Time Frame: Baseline, 6 Months
Population: Enrolled participants who completed assessments on their sexual risk behaviors (e.g. condomless anal sex (CAS) acts) at baseline and 6 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 445 | 454
Participants
  Baseline | 304 | 312
  6 Month Follow-up: number analyzed (Participants) | 340 | 380
  6 Month Follow-up | 133 | 156
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Superiority; p = 0.60, Regression, Logistic; Prevalence Ratio = 0.95, 95% CI 2-sided [0.80 to 1.14]

3. Primary Outcome: Participants Self-Reporting Condomless Anal Sex at Baseline and 12 Months
Description: Change in self-report of condomless anal sex acts at twelve months.
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on their sexual risk behaviors (e.g. condomless anal sex (CAS) acts) at baseline and 12 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 445 | 454
Participants
  Baseline | 304 | 312
  12 Month Follow-up: number analyzed (Participants) | 366 | 391
  12 Month Follow-up | 136 | 173
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Superiority; p = 0.04, Regression, Logistic; Prevalence Ratio = 0.83, 95% CI 2-sided [0.70 to 0.99]

4. Primary Outcome: Number of Participants With Occurrence of Sexually Transmitted Infections (STIs) at Baseline
Description: The incidence (number of new cases or diagnoses) of chlamydia and gonorrhea at baseline.
Time Frame: Baseline
Population: Enrolled participants who returned STI test kits for analysis at baseline. Denominator varies by testing site and study arm: urethral (control - 452; intervention - 441) rectal (control - 449; intervention - 442)
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 443 | 453
Participants
  Urethral Chlamydia: number analyzed (Participants) | 441 | 452
  Urethral Chlamydia | 15 | 7
  Urethral Gonorrhea: number analyzed (Participants) | 441 | 452
  Urethral Gonorrhea | 3 | 4
  Rectal Chlamydia: number analyzed (Participants) | 442 | 449
  Rectal Chlamydia | 47 | 30
  Rectal Gonorrhea: number analyzed (Participants) | 442 | 449
  Rectal Gonorrhea | 29 | 16
  Any STI | 82 | 50

5. Primary Outcome: Number of Participants With Occurrence of Sexually Transmitted Infections (STIs) at 12 Months
Description: The incidence (number of new cases or diagnoses) of chlamydia and gonorrhea at twelve months.
Time Frame: 12 months
Population: Enrolled participants who returned STI test kits for analysis at 12 month follow-up.
  Denominator varies by testing site and study arm: urethral (control - 374; intervention - 359) rectal (control - 374; intervention - 356)
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 359 | 374
Participants
  Urethral Chlamydia | 4 | 7
  Urethral Gonorrhea | 1 | 3
  Rectal Chlamydia: number analyzed (Participants) | 356 | 374
  Rectal Chlamydia | 22 | 38
  Rectal Gonorrhea: number analyzed (Participants) | 356 | 374
  Rectal Gonorrhea | 13 | 15
  Any STI | 31 | 54
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Superiority; p = 0.01, Z-test; Risk Ratio (RR) = 0.60, 95% CI 2-sided [0.38 to 0.95]

6. Secondary Outcome: Mean Score of Condom Errors at Baseline and 3 Months
Description: The change in frequency that a participant has not correctly used a condom (for example, starting sex without a condom or using the wrong lube with condoms) at three months. Must have reported anal sex and using a condom with a partner at both time points. Range of scores - 0-11; higher scores = more errors.
Time Frame: Baseline, 3 Months
Population: Enrolled participants who completed assessments on condom errors at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 140 | 150
units on a scale
  Baseline | 4.28 (2.16) | 4.05 (2.12)
  3 Month Follow-up | 3.23 (2.27) | 3.45 (2.09)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.150, Regression, Linear

7. Secondary Outcome: Percentage of Correct Responses on HIV Knowledge Assessment at Baseline and 3 Months
Description: The change in number of HIV statements (e.g. "Only the receptive/bottom partner is at risk of being infected with HIV during anal sex", "There is a vaccine that can stop people from getting HIV", and "A natural skin (lamb skin) condom works better against HIV than does a latex condom") correctly labeled as true or false at three months. All 26 statements were recoded such that correct responses = 1 and incorrect or 'don't know' responses = 0. Composite scores were calculated to reflect the percentage of correct responses. Higher scores reflect greater knowledge of HIV transmission/risk.
Time Frame: Baseline, 3 Months
Population: Enrolled participants who completed assessments on HIV knowledge at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 348 | 409
percentage of correct responses
  Baseline | 85.93 (13.00) | 86.41 (11.64)
  3 Month Follow-up | 89.11 (11.22) | 88.68 (11.80)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.374, Regression, Linear

8. Secondary Outcome: Mean Score of Motivation and Behavioral Skills at Baseline and 3 Months
Description: At three months, the change in:
  * Motivation (for example, intentions to use condoms, perceived threat of HIV or STI infection, desire to become safer)
  * Social Norms (for example, partners, friends, or family members opinions about condom use)
  * Behavioral Skills (for example, negotiating condom use)
  Motivational Self-Rating - higher score = higher motivation; range 1-4 Social Norms - higher score = higher endorsement of social norms; range 1-5 Behavioral Skills - higher score = less perceived difficulty using condoms; range 1-4
Time Frame: Baseline, 3 Months
Population: Enrolled participants who completed assessments on motivation & behavioral skills at baseline and 3 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 348 | 409
units on a scale
  Baseline - Motivational Self-Rating | 3.11 (0.80) | 3.02 (0.87)
  3 Month Follow-up - Motivational Self-Rating | 3.11 (0.91) | 3.03 (0.92)
  Baseline - Social Norms | 4.36 (0.54) | 4.33 (0.53)
  3 Month Follow-up - Social Norms | 4.37 (0.62) | 4.32 (0.62)
  Baseline - Behavioral Skills | 1.36 (0.39) | 1.39 (0.39)
  3 Month Follow-up - Behavioral Skills | 1.28 (0.35) | 1.38 (0.42)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Motivation items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.919, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Social Norms items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.493, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Behavioral Skills items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.002, Regression, Linear

9. Secondary Outcome: Mean Score of Health Protective Communication Skills at Baseline and 3 Months
Description: The change in how frequently health protection (for example, condom use and regular HIV testing) is discussed with sex partners at three months. Higher score = less HPC skills; range 1-4 for each item on scale (relationship maintenance, condom use, and HIV testing).
Time Frame: Baseline, 3 Months
Population: Enrolled participants who completed assessments on health protective communication (HPC) Relationship & condom items: must have reported vaginal/anal sex partner in prev. 3 months at both time points HIV testing items: must have reported NEW vaginal/anal sex partner in prev. 3 months at both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 236 | 292
units on a scale
  Baseline - HPC Relationship Maintenance | 1.34 (0.75) | 1.36 (0.80)
  3 Month Follow-up - HPC Relationship Maintenance | 1.46 (0.89) | 1.37 (0.83)
  Baseline - HPC Condom Use | 1.32 (0.86) | 1.10 (0.81)
  3 Month Follow-up - HPC Condom Use | 1.38 (0.92) | 1.22 (0.97)
  Baseline - HPC HIV Testing: number analyzed (Participants) | 63 | 74
  Baseline - HPC HIV Testing | 0.76 (0.75) | 0.43 (0.63)
  3 Month Follow-up - HPC HIV Testing: number analyzed (Participants) | 63 | 74
  3 Month Follow-up - HPC HIV Testing | 0.71 (0.73) | 0.61 (0.63)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Relationship Maintenance items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.067, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Condom Use items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.135, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for HIV Testing items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.025, Regression, Linear

10. Secondary Outcome: Number of Participants Reporting Drug Use Before Sex at Baseline and 12 Months
Description: The change in number of participants who report using illegal drugs or drugs not prescribed by a doctor before sex.
Time Frame: Baseline, 12 Month
Population: Enrolled participants who completed assessments on drug use before sex at baseline and 12 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 370 | 392
Participants
  Baseline | 100 | 108
  12 Month Follow-up | 92 | 84
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.138, Regression, Logistic

11. Secondary Outcome: Mean Score of Condom Errors at Baseline and 6 Months
Description: The change in frequency that a participant has not correctly used a condom (for example, starting sex without a condom or using the wrong lube with condoms) at six months. Must have reported anal sex and using a condom with a partner at both time points. Range of scores - 0-11; higher scores = more errors
Time Frame: Baseline, 6 Months
Population: Enrolled participants who completed assessments on condom errors at baseline and 6 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 124 | 121
units on a scale
  Baseline | 4.29 (2.14) | 3.96 (2.13)
  6 Month Follow-up | 3.09 (2.20) | 3.12 (2.35)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.173, Regression, Linear

12. Secondary Outcome: Percentage of Correct Responses on HIV Knowledge Assessment at Baseline and 6 Months
Description: The change in number of HIV statements (e.g. "Only the receptive/bottom partner is at risk of being infected with HIV during anal sex", "There is a vaccine that can stop people from getting HIV", and "A natural skin (lamb skin) condom works better against HIV than does a latex condom") correctly labeled as true or false at six months. All 26 statements were recoded such that correct responses = 1 and incorrect or 'don't know' responses = 0. Composite scores were calculated to reflect the percentage of correct responses. Higher scores reflect greater knowledge of HIV transmission/risk.
Time Frame: Baseline, 6 Months
Population: Enrolled participants who completed assessments on HIV Knowledge at baseline and 6 month.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 342 | 380
percentage of correct responses
  Baseline | 85.78 (13.21) | 86.69 (11.59)
  6 Month Follow-up | 88.96 (12.52) | 89.25 (12.31)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.567, Regression, Linear

13. Secondary Outcome: Mean Score of Motivation and Behavioral Skills at Baseline and 6 Months
Description: At six months, the change in:
  * Motivation (for example, intentions to use condoms, perceived threat of HIV or STI infection, desire to become safer)
  * Social Norms (for example, partners, friends, or family members opinions about condom use)
  * Behavioral Skills (for example, negotiating condom use)
  Motivational Self-Rating - higher score = higher motivation; range 1-4 Social Norms - higher score = higher endorsement of social norms; range 1-5 Behavioral Skills - higher score = less perceived difficulty using condoms; range 1-4
Time Frame: Baseline, 6 Months
Population: Enrolled participants who completed assessments on motivation & behavioral skills at baseline and 6 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 342 | 380
units on a scale
  Baseline - Motivational Self-Rating | 3.13 (0.80) | 3.03 (0.85)
  6 Month Follow-up - Motivational Self-Rating | 3.12 (0.90) | 3.04 (0.93)
  Baseline - Social Norms | 4.35 (0.54) | 4.34 (0.53)
  6 Month Follow-up - Social Norms | 4.31 (0.66) | 4.27 (0.72)
  Baseline - Behavioral Skills | 1.36 (0.39) | 1.39 (0.38)
  6 Month Follow-up - Behavioral Skills | 1.30 (0.40) | 1.37 (0.41)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for motivation items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.861, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for social norms items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.628, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for behavioral skills items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.151, Regression, Linear

14. Secondary Outcome: Mean Score of Health Protective Communication Skills at Baseline and 6 Months
Description: The change in how frequently health protection (for example, condom use and regular HIV testing) is discussed with sex partners at six months. Higher score = less HPC skills; range 1-4 for each item on scale (relationship maintenance, condom use, and HIV testing).
Time Frame: Baseline, 6 Months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 221 | 256
units on a scale
  Baseline - HPC Relationship Maintenance | 1.36 (0.75) | 1.35 (0.78)
  6 Month Follow-up - HPC Relationship Maintenance | 1.65 (0.91) | 1.39 (0.83)
  Baseline - HPC Condom Use | 1.35 (0.85) | 1.06 (0.78)
  6 Month Follow-up - HPC Condom Use | 1.25 (0.95) | 1.10 (0.96)
  Baseline - HPC HIV Testing: number analyzed (Participants) | 56 | 72
  Baseline - HPC HIV Testing | 0.61 (0.68) | 0.48 (0.70)
  6 Month Follow-up - HPC HIV Testing: number analyzed (Participants) | 56 | 72
  6 Month Follow-up - HPC HIV Testing | 0.74 (0.88) | 0.69 (0.80)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Relationship Maintenance items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.001, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Condom Use items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.067, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for HIV Testing items; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.637, Regression, Linear

15. Secondary Outcome: Mean Score of Condom Errors at Baseline and 12 Months
Description: The change in frequency that a participant has not correctly used a condom (for example, starting sex without a condom or using the wrong lube with condoms) at twelve months. Must have reported anal sex and using a condom with a partner at both time points. Range of scores - 0-11; higher scores = more errors.
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on their condom errors at baseline and 12 month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 112 | 115
units on a scale
  Baseline | 4.31 (2.31) | 4.02 (2.23)
  12 Month Follow-up | 3.30 (2.49) | 3.16 (2.24)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.862, Regression, Linear

16. Secondary Outcome: Percentage of Correct Responses on HIV Knowledge Assessment at Baseline and 12 Months
Description: The change in number of HIV statements (e.g. "Only the receptive/bottom partner is at risk of being infected with HIV during anal sex", "There is a vaccine that can stop people from getting HIV", and "A natural skin (lamb skin) condom works better against HIV than does a latex condom") correctly labeled as true or false at twelve months. All 26 statements were recoded such that correct responses = 1 and incorrect or 'don't know' responses = 0. Composite scores were calculated to reflect the percentage of correct responses. Higher scores reflect greater knowledge of HIV transmission/risk.
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on their HIV Knowledge at baseline and 12 month follow-up.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 370 | 392
percentage of correct responses
  Baseline | 85.02 (13.67) | 86.76 (10.88)
  12 Month Follow-up | 88.46 (13.15) | 89.94 (10.34)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Other — Generalized Linear Mixed Model statistical test used; p = 0.762, Regression, Linear

17. Secondary Outcome: Mean Score of Motivation and Behavioral Skills at Baseline and 12 Months
Description: At twelve months, the change in:
  * Motivation (for example, intentions to use condoms, perceived threat of HIV or STI infection, desire to become safer)
  * Social Norms (for example, partners, friends, or family members opinions about condom use)
  * Behavioral Skills (for example, negotiating condom use)
  Motivational Self-Rating - higher score = higher motivation; range 1-4 Social Norms - higher score = higher endorsement of social norms; range 1-5 Behavioral Skills - higher score = less perceived difficulty using condoms; range 1-4
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on motivation & behavioral skills at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 370 | 392
units on a scale
  Baseline - Motivational Self-Rating | 3.13 (0.80) | 3.02 (0.87)
  12 Month Follow-up - Motivational Self-Rating | 2.93 (0.94) | 2.97 (0.99)
  Baseline - Social Norms | 4.32 (0.58) | 4.34 (0.53)
  12 Month Follow-up - Social Norms | 4.24 (0.65) | 4.23 (0.67)
  Baseline - Behavioral Skills | 1.35 (0.39) | 1.39 (0.38)
  12 Month Follow-up - Behavioral Skills | 1.38 (0.47) | 1.39 (0.46)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Motivation items; Test type: Superiority; p = 0.043, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Social Norm items; Test type: Superiority; p = 0.617, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Behavioral Skills items; Test type: Superiority; p = 0.570, Regression, Linear

18. Secondary Outcome: Mean Score of Health Protective Communication Skills at Baseline and 12 Months
Description: The change in how frequently health protection (for example, condom use and regular HIV testing) is discussed with sex partners at twelve months. Higher score = less HPC skills; range 1-4 for each item on scale (relationship maintenance, condom use, and HIV testing).
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on health protective communication (HPC) Relationship & condom items: must have reported vaginal/anal sex partner in prev. 3 months at both time points HIV testing items: must have reported NEW vaginal/anal sex partner in prev. 3 months at both time points Higher score = less HPC skills; range 1-4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 245 | 284
units on a scale
  Baseline - HPC Relationship Maintenance | 1.32 (0.79) | 1.31 (0.80)
  12 Month Follow-up - HPC Relationship Maintenance | 1.65 (0.88) | 1.45 (0.87)
  Baseline - HPC Condom Use | 1.32 (0.83) | 1.09 (0.85)
  12 Month Follow-up - HPC Condom Use | 1.12 (0.95) | 0.96 (0.89)
  Baseline - HPC HIV Testing: number analyzed (Participants) | 52 | 74
  Baseline - HPC HIV Testing | 0.57 (0.68) | 0.48 (0.65)
  12 Month Follow-up - HPC HIV Testing: number analyzed (Participants) | 52 | 74
  12 Month Follow-up - HPC HIV Testing | 0.64 (0.73) | 0.56 (0.68)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Relationship Maintenance items; Test type: Superiority; p = 0.036, Regression, Linear
Statistical Analysis 2: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for Condom Use items; Test type: Superiority; p = 0.837, Regression, Linear
Statistical Analysis 3: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Analysis for HIV Testing items; Test type: Superiority; p = 0.953, Regression, Linear

19. Secondary Outcome: Mean Score of Feelings of HIV Invulnerability at Baseline and 12 Months
Description: The change in effect that HIV testing has on health beliefs (for example, "I cannot get HIV") and sexual behaviors at twelve months. Range 1-5; higher scores = more feelings of invulnerability
Time Frame: Baseline, 12 Months
Population: Enrolled participants who completed assessments on HIV invulnerability at baseline and 12 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 370 | 392
units on a scale
  Baseline | 1.92 (0.75) | 1.84 (0.74)
  12 Month Follow-up | 2.05 (0.78) | 1.95 (0.74)
Statistical Analysis 1: Comparison: Keep It Up! Intervention vs HIV Knowledge Control; Test type: Superiority; p = 0.719, Regression, Linear

20. Other Pre Specified Outcome: Participant Rating of Intervention Acceptability and Tolerability
Description: Participant rating of how much they enjoyed the intervention and participant feedback and suggestions for improvement. Range 1-4; higher scores indicate greater acceptability.
Time Frame: Immediately following completion of intervention (up to 3 weeks after intervention is started by participant)
Population: Enrolled participants who completed assessments on intervention acceptability immediately following completion of intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 375 | 434
units on a scale | 3.52 (0.41) | 3.50 (0.41)

21. Other Pre Specified Outcome: Participant Location
Description: Log of where participants completed the intervention sessions (participants can select multiple locations).
Time Frame: Immediately following completion of intervention (up to 3 weeks after intervention is started by participant)
Population: Participants who reported information about the locations where they completed the intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 375 | 434
Participants
  At Home, Not in Bedroom | 183 | 213
  At Home, In Bedroom | 231 | 303
  Coffee Shop | 21 | 29
  Community Center | 16 | 13
  Library | 25 | 36
  Friend's House | 32 | 36
  Other | 69 | 105

22. Other Pre Specified Outcome: Participant Experiences of Harm at 3 Month Follow-up
Description: Log of any negative experiences or harm experienced by participant at three months.
Time Frame: 3 Months
Population: Number of participants who reported negative health experiences at 3 Month Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 348 | 409
Participants | 0 | 0

23. Other Pre Specified Outcome: Participant Experiences of Harm at 6 Month Follow-up
Description: Log of any negative experiences or harm experienced by participant at six months.
Time Frame: 6 Months
Population: Number of participants who reported negative health experiences at 6 Month Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 342 | 380
Participants | 0 | 0

24. Other Pre Specified Outcome: Participant Experiences of Harm at 12 Month Follow-up
Description: Log of any negative experiences or harm experienced by participant at twelve months.
Time Frame: 12 Months
Population: Number of participants who reported negative health experiences at 12 Month Follow-up as a result of participating in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 370 | 392
Participants | 0 | 0

25. Other Pre Specified Outcome: Occurrence of Sexually Transmitted Infections (STIs) at 3 Months
Description: The incidence (number of new cases or diagnoses) of chlamydia and gonorrhea at 3 month follow-up. Only measured for participants who initially tested positive for chlamydia or gonorrhea at baseline.
Time Frame: 3 Months
Population: Participants who were positive for an STI at baseline, were sent a follow-up test kit at 3 Month Follow-up, and tested positive again.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 55 | 32
Participants
  Urethral Chlamydia | 1 | 1
  Urethral Gonorrhea | 0 | 0
  Rectal Chlamydia | 12 | 11
  Rectal Gonorrhea | 6 | 4
  Any STI | 9 | 5

26. Other Pre Specified Outcome: Occurrence of Sexually Transmitted Infections (STIs) at 6 Months
Description: The incidence (number of new cases or diagnoses) of chlamydia and gonorrhea at 6 month follow-up. Only measured for participants who initially tested positive for chlamydia or gonorrhea at baseline.
Time Frame: 6 Months
Population: Participants who were positive for an STI at baseline, were sent a follow-up test kit at 6 Month Follow-up, and tested positive again.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 50 | 26
Participants
  Urethral Chlamydia | 0 | 0
  Urethral Gonorrhea | 0 | 0
  Rectal Chlamydia | 7 | 5
  Rectal Gonorrhea | 2 | 0
  Any STI | 9 | 5

27. Other Pre Specified Outcome: Level of Privacy
Description: Log of the levels of privacy of the locations where participants completed intervention.
Time Frame: Immediately following completion of intervention (up to 3 weeks after intervention is started by participant)
Population: Participants who reported information about the locations where they completed the intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
Number analyzed (Participants) | 373 | 433
Participants
  Not Private At All | 14 | 28
  Somewhat Private | 74 | 100
  Moderately Private | 81 | 106
  Completely Private | 204 | 199

ADVERSE EVENTS:
Time Frame: Adverse event data collected for nearly 4 years (May 2013 - March 2017)
Description: The adverse events that are reported differ from the clinicaltrials.gov definitions.
  Serious Non-compliance: Failure to follow the regulations, requirements and/or determinations of the IRB that adversely affects the rights or welfare of subjects.
  UPIRSO: Any incident that meets ALL of the following conditions:
  1. unexpected
  2. related or possibly related to participation in the research
  3. suggests that the research places human subjects or others at a greater risk of harm
Arm/Group | Keep It Up! Intervention | HIV Knowledge Control
All-Cause Mortality (participants affected / at risk) | 0/445 | 0/456
Serious Adverse Events (participants affected / at risk) | 11/445 | 13/456
Other Adverse Events (participants affected / at risk) | 0/445 | 0/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keep It Up! Intervention (N=445) | HIV Knowledge Control (N=456)
Confidentiality Breach 3.27.14 (Social circumstances) | 10 (10) | 12 (12) — On March 27, 2014, a group email was sent to study participants using the carbon copy (cc:) field instead of blind carbon copy (bcc:) field. IRB determined to be a UPIRSO.
Confidentiality Breach 9.11.15 (Social circumstances) | 1 (1) | 1 (1) — On September 11, 2015, a study participant received an email from a project research assistant that contained the assessment login information and email address of another participant. IRB determined to be serious non-compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT01836445/Prot_001.pdf
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT01836445/SAP_002.pdf
  • Informed Consent Form (2014-11-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT01836445/ICF_000.pdf